CLINICAL TRIAL: NCT03819595
Title: "BIZI ORAIN": Exercise for All People With Cancer
Brief Title: BIZI ORAIN: Exercise for All People With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Nere Mendizabal, Principal Investigator, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 18/00929
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-07

CONDITIONS: Cancer; Quality of Life; Functional Capacity; Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised arm (Experimental): Supervised exercise. The intervention will be a free 12-week, small-group (~10 people) exercise program supervised by specially trained instructors, combining two weekly 1h sessions of moderate to high intensity aerobic and strength exercise. Participants are encouraged to undertake an additional group-based walking exercise guided by target heart rates.
  Interventions: Other: Supervised exercise
- Control arm (Active Comparator): Supervised exercise.The intervention will be a Personalized program (PVS), of proven effectiveness for the promotion of physical activity, diet and smoking cessation.
  After 3 months, it become supervised arm
  Interventions: Other: Supervised exercise; Other: Personalized Program PVS

INTERVENTIONS:
Other: Supervised exercise — a free 12-week, small-group (~10 people) exercise program supervised by specially trained instructors, combining two weekly 1h sessions of moderate to high intensity aerobic and strength exercise. Participants are encouraged to undertake an additional group-based walking exercise guided by target heart rates.
Other: Personalized Program PVS — a standardized promotion prescription of physical activity, balanced diet and smoking cessation, using the computer tool "Promote Healthy Living" integrated into the electronic medical record.
  Arms: Control arm

SUMMARY:
Background: Physical exercise should be an essential component of the therapeutic plan for every person diagnosed with cancer. However, most of these patients are inactive and only a few of them receive prescription and follow-up for safe and effective exercise plans.

Objective: in a first experimental phase, we will evaluate actual implementation (reach and adherence) and clinical effectiveness (physical fitness, quality of life and symptoms) of the BIZI ORAIN (BO) exercise program, for all patients diagnosed with cancer, compared to standardized physical activity counseling. In a second, observational phase, we will evaluate the association between levels of physical activity actually performed by all the participants and their 12 months evolution, in terms of physical fitness, quality of life, symptomatology and survival.

Design: Hybrid study, with a first experimental phase in which patients diagnosed with cancer will be randomly assigned to two parallel groups, one that immediately performs the BO program for 12 weeks and the other one that performs the same programme three months later (delayed treatment). In the second phase, observational, the entire cohort of participants will be followed-up for one year. Population: Any person diagnosed with cancer in the previous two years (minimum sample size = 1013) free of bone metastases, hematological or other exercise contraindications.

BIZI ORAIN program: based on the "Life Now" program of the Australian Cancer Council, BO is a 12-week small-group exercise program supervised by specially trained instructors combining moderate to high intensity aerobic and strength exercises (three 1 hour sessions a week).

Outcome measurements: the main outcome variable will be the change in functional capacity at three months (400 meters walk test). Secondary variables include mortality, quality of life (general SF-36 and cancer specific quality of life -European Organization for Research and Treatment of Cancer QLQ-C-30-), symptoms (Cancer-related fatigue - Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue), exposure to physical activity level objectively registered with Actigraph wGT3X-BT accelerometer, chronic inflammation (C-reactive protein, adiponectin, and pro-inflammatory cytokines Il-1, Il-6 , and TNF-), body composition and bone health (dual-energy X-ray absorptiometry), measured at 0, 3, 6, and 12 months.

Analyses: changes observed in the outcome variables at three months will be compared between patients assigned to BO and to the reference group (delayed treatment) using analysis of the covariance, adjusted for baseline levels. To analyze the association between over time change in physical activity and the outcome variables mixed effects longitudinal models will be used for repeated measures throughout the 12 months of follow-up. Cox proportional hazards models will be used for the survival analysis. Qualitative analyses will combine a deductive approach with an inductive one based on Grounded Theory. In the deductive approach, the researchers will identify several thematic categories related to the Consolidated Framework for Implementation Research. Conclusions: BO is the first experience in Spain of a population-based exercise program that will guarantee, through a scientific evaluation, both clinical and implementation results. This will drastically advance the treatment of people suffering from cancer helping them to reverse the effects of their disease, the adverse effects of the therapies and to improve anti-cancer treatment efficacy, their quality of life and survival

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with cancer within the previous 2 years, under treatment or finished

Exclusion Criteria:

* Neutropenia
* severe anemia
* bone metastases
* any musculoskeletal, cardiovascular or neurological disorder that could place the participant at risk of injury or illness resulting from the exercise program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Change in Functional Capacity (400 meters walk test) | One year follow up. Measures at 0,3,6 and 12 months
  The 400 meters walk Test applies to assess functional capacity, as well as a predictor of morbidity and mortality in people with different pathologies. Most of the daily activities that the patients with these pathologies are performed at submaximal exercise intensity, similar to this test is performed. It would be measured at 0, 3,6 and 12 months.

SECONDARY OUTCOMES:
Change in Quality of life (general SF-36) | 1 year follow up. Measures at 0,3,6 and 12 months
  The HRQL questionnaire is measured blindly with self-administered questionnaires: the Spanish version of the SF-36 and. Questionnaire will be filled out before and after the intervention. SF-36 generates an 8-dimension health profile and two summary scores for the physical and mental components. This questionnaire has been validated in the Spanish population. Measured at 0, 3, 6 and 12 months.
Change in Quality of life (cancer specific quality of life -European Organization for Research and Treatment of Cancer QLQ-C-30) | 1 year follow up. Measures at 0,3,6 and 12 months
  Cancer specific quality of life is evaluated by the European Organisation for Research and Treatment of Cancer (QLQ-C-30) questionnaire (Aaronson et al., 1993). The QLQ-C-30 questionnaire includes five functional domains (physical, role, cognitive, emotional and social; higher scores represent greater function/quality of life) and three symptom scales (fatigue, pain and nausea; lower scores represent greater quality of life/less symptom severity).Measured at 0, 3, 6 and 12 months
symptoms (Cancer-related fatigue - Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | 1 year follow up. Measures at 0,3,6 and 12 months
  a 13 items scale that measures the cancer related fatigue. The FACT-G scoring guide identifies those items that must be reversed before being added to obtain subscale totals. Negatively stated items are reversed by subtracting the response from "4". After reversing proper items, all subscale items are summed to a total, which is the subscale score.The higher score the score, the better the QOL. Measured at 0, 3, 6 and 12 months
physical activity level | 1 year follow up. Measures at 0,3,6 and 12 months
  objectively registered with Actigraph wGT3X-BT accelerometer. Measured at 0, 3, 6 and 12 months
concentration of Lipids | 3 months. Measures at 0,3 months.
  Lipids:cholesterol (mg/dl), tryglicerides (mg/dl), HDL (mg/dl), LDL(mg/dl). Measured at baseline, and 3 months
concentration of C reactive protein | 3 months. Measures at 0,3 months.
  C reactive protein (mg/l). Measured at 0, and 3 months
concentration of glucose | 3 months. Measures at 0,3 months.
  glycemia (mg/dl). Measured at 0, and 3 months
concentration of Insulin | 3 months. Measures at 0,3 months.
  Insulin (microU/ml). Measured at 0, and 3 months
concentration of adiponectin | 3 months. Measures at 0,3 months.
  Exercise specific parameters: adiponectin (microgr/mL). Measured at baseline, and 3 months
concentration of TNF | 3 months. Measures at 0,3 months.
  Exercise specific parameters: TNF in Cancer patients (pg/ml) .Measured at baseline, and 3 months
concentration of Interleukins II-1 and II-6 | 3 months. Measures at 0,3 months.
  Exercise specific parameters: Interleukins II-1 and II-6 (pg/ml). Measured at baseline, and 3 months
Change in Body composition (fat and muscular weight). (BMI) | 1 year follow up. Measures at 0,3,6 and 12 months
  Body Mass Index (BMI): Diagnoses and classifies obesity. weight and height will be combined to report BMI in kg/m^2). Measured at baseline, and 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nere Mendizabal, Principal Investigator — Basque Health Service
Locations (1):
- Primary care research unit of Bizkaia, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arietaleanizbeaskoa MS, Gil Rey E, Mendizabal Gallastegui N, Garcia-Alvarez A, De La Fuente I, Dominguez-Martinez S, Pablo S, Coca A, Gutierrez Santamaria B, Grandes G. Implementing Exercise in Standard Cancer Care (Bizi Orain Hybrid Exercise Program): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Aug 9;10(8):e24835. doi: 10.2196/24835. PMID 34383676